CLINICAL TRIAL: NCT06718218
Title: A Combination Mindfulness and Music Intervention for Acute Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00004916_BB
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pain; Acute Pain
Keywords: Mindfulness
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness Pain Management (Active Comparator)
  Interventions: Behavioral: Mindfulness Pain Management
- Mindfulness Recording With Sustained Tone (Experimental)
  Interventions: Behavioral: Mindfulness Recording With Sustained Tone
- Mindfulness Recording with Binaural Beats (Experimental)
  Interventions: Behavioral: Mindfulness Recording with Binaural Beats
- Mindfulness Recording with Binaural Beats and Theta Music (Experimental)
  Interventions: Behavioral: Mindfulness Recording with Binaural Beats and Theta Music

INTERVENTIONS:
Behavioral: Mindfulness Pain Management — Participants will listen to a 5-minute audio recording of a mindfulness exercise consisting of a 1-minute introduction to mindful pain management and a 4-minute mindfulness practice.
  Arms: Mindfulness Pain Management
Behavioral: Mindfulness Recording With Sustained Tone — Participants will listen to a 5-minute audio recording of a mindfulness exercise consisting of a 1-minute introduction to mindful pain management and a 4-minute mindfulness practice, that is accompanied by a sustained low C tone at 65.41 Hertz.
  Arms: Mindfulness Recording With Sustained Tone
Behavioral: Mindfulness Recording with Binaural Beats — Participants will listen to a 5-minute audio recording of a mindfulness exercise consisting of a 1-minute introduction to mindful pain management and a 4-minute mindfulness practice that is accompanied by binaural beats resulting from the delivery of a sustained 65.41 Hertz tone in the left ear and a sustained 69.41 Hertz tone in the right ear.
  Arms: Mindfulness Recording with Binaural Beats
Behavioral: Mindfulness Recording with Binaural Beats and Theta Music — Participants will listen to a 5-minute audio recording of a mindfulness exercise consisting of a 1-minute introduction to mindful pain management and a 4-minute mindfulness practice that is accompanied by binaural beats resulting from the delivery of a sustained 65.41 Hertz tone in the left ear and a sustained 69.41 Hertz tone in the right ear as well as instrumental theta wave music.
  Arms: Mindfulness Recording with Binaural Beats and Theta Music

SUMMARY:
This project is a single-site, four-arm, randomized controlled trial evaluating a combination mindfulness + music intervention on acute pain among patients in an orthopedic clinic waiting room. Participants will be randomized to one of four conditions: 1) a 5-minute mindfulness recording, 2) a 5-minute mindfulness recording with an accompanying sustained tone at 65.41 Hertz, 3) a 5-minute mindfulness recording with an accompanying binaural beat set at 65.41 Hertz in the left ear and 69.41 Hertz in the right ear, or 4) a 5-minute mindfulness recording with an accompanying binaural beat set at 65.41 Hertz in the left ear and 69.41 Hertz in the right ear as well as instrumental, theta wave music.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Receiving pain treatment at Tallahassee Orthopedic Center
* Understanding English instructions fluently

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before and after 5-minute audio recording
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before and after 5-minute audio recording
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Change in Anxiety Numeric Rating Scale | Immediately before and after 5-minute audio recording
  Change in anxiety from baseline will be assessed with an item adapted from the Generalized Anxiety Disorder 2-item. Scores range from 0 to 10, with higher scores reflecting greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No